CLINICAL TRIAL: NCT03506464
Title: Short-term Effects of a Myofascial Release on Elasticity in Patients With Plantar Fasciitis: A Pre-post Evaluation With Sonoelastography
Brief Title: Myofascial Release in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, María Elena del Baño-Aledo, Principal Investigator, Universidad de Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sono2018
Record Dates: First submitted 2018-02-19; First posted 2018-04-24 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fasciitis; physical therapy; sonoelastography
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Myofascial Release Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plantar fasciitis group (Experimental): Myofascial release technique
  Interventions: Procedure: Myofascial Release Technique
- control group (No Intervention): None of the control group received the treatment

INTERVENTIONS:
Procedure: Myofascial Release Technique — The same described in the arm description
  Arms: plantar fasciitis group

SUMMARY:
Background: Plantar fasciitis is the most common cause of heel pain in runners. No studies have described the short-term effects of myofascial release on plantar fasciitis using ultrasound.

Objectives: To describe the immediate sonoelastographic changes in the plantar fascia of amateur runners with fasciitis after applying a myofascial release technique.

Design: A single-centre, experimental and controlled study.

Method: Patients with plantar fasciitis and a group of healthy subjects will be examined using B-mode and real time sonoelastography scanning. Fascia thickness, echointensity and echovariation of the color histogram will be analyzed pre- and post intervention. A two-way (Group × Time) repeated measures ANOVA will be performed.

DETAILED DESCRIPTION:
Participants

Subjects of the plantar fasciitis group (PFG) will be recruited in May2018 to apply to them a myofascial release technique.

Healthy volunteers without a history of plantar fascia disease will be recruited as control group (CG).

The examination will be included B-mode scanning and real time sonoelastography using an US scanner with linear array transducer (ML6-15). All examinations will be conducted by a sonographer with more than 10 years' experience in musculoskeletal imaging.

Using a standardized protocol three images of every pre-post intervention video will be stored uncompressed and with no losses in bitmap format (bmp), and the mean value of the histogram components will be used for statistical analysis. The examination protocol shows good reliability, and has been reported previously.

ImageJ 1.45 software will be used to perform quantitative analysis of gray-scale images and the color histogram of the elastogram.

ELIGIBILITY:
Inclusion Criteria:

* heel pain at the proximal fascia insertion
* worse pain when waking up in the morning or after a period of rest
* a visual analog score (VAS) of more than 4 on a scale of 10

Exclusion Criteria:

* Patients who had undergone surgery or steroid injections to the heel will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Changes in thickness of the plantar fascia | Measured twice. pre and post treatment. Post treatment examination will be carried out 10 minutes after the intervention concludes.
  Measured from the anterior edge of the inferior calcaneal border vertically to the inferior border of the plantar fascia
Changes in echointensity | Measured twice. pre and post treatment. Post treatment examination will be carried out 10 minutes after the intervention concludes.
  The EI of the color histogram computed the mean value of intensity of red, green and blue channels (color intensity range, 0-255) within a given area
Changes in Echovariation | Measured twice. pre and post treatment. Post treatment examination will be carried out 10 minutes after the intervention concludes.
  Determined as the relation between standard deviation and mean of pixel intensity obtained from the histogram

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena del Baño-Aledo, Dr, Principal Investigator — Universidad de Murcia
Locations (1):
- María Elena del Baño Aledo, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No